CLINICAL TRIAL: NCT05351814
Title: The Effect Of Core Stabilization Exercises In Patellofemoral Pain Syndrome
Brief Title: Effectiveness Of Core Stabilization Exercises In Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Ceren Demirtaş, PHYSIOTHERAPIST, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-128
Record Dates: First submitted 2022-04-04; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Core Stability; Patellofemoral Pain; Exercise Therapy; Core Balance; Flexibility
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Individuals will be divided into two groups by computerized randomization. Control group; Traditional patellofemoral pain syndrome exercises, (n=20) Core stability group; Core stabilization and hip exercises will be given in addition to traditional patellofemoral pain syndrome exercises. (n=20)
Who Masked: Participant
Masking Description: Individuals will be divided into two groups by computerized randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group; traditional patellofemoral pain syndrome exercises; isometric exercises 3 sets of 10 repetitions in one session, balance exercise 30/45 sec, one leg balance exercise 45/60 sec , stretching exercises 4 sets 5 repetitions 20 sec duration, off kinetic chain (CHC) AND open kinetic chain (ACZ) exercises were planned as 3 sets for 4 weeks and 3 days a week.
  Interventions: Other: Exercise
- Core Stability group (Experimental): Core stability group; In addition to traditional patellofemoral pain syndrome exercises; hip muscle strengthening exercises are 3 sets of 10 repetitions in each session, and (core) stabilization exercises are 1st and 2nd weeks 2 sets 15 repetitions 3rd and 4th weeks 2 sets 5 repetition was planned for 4 weeks and 3 days a week.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — While the patients will be exercised with a physiotherapist 1 day a week, the treatment will be followed as a home exercise program 2 days a week.

SUMMARY:
The aim of this randomized controlled study; To investigate the multifactorial effectiveness of core stabilization exercises applied in patients diagnosed with patellofemoral pain syndrome.

20/60 years old/with retropatellar pain that occurs during at least two of the activities and persists for at least one month While patients diagnosed with patellofemoral pain syndrome (PFPS) were included in the study; Patients with meniscus and ligament lesions, osteoarthritis, patellofemoral dislocation and/or subluxation history, osseous anomalies and history of knee surgery, pregnancy status, and patients using analgesics and anti-inflammatory drugs will not be included in the study.

Individuals will be divided into two groups by computerized randomization. Control group; Traditional patellofemoral pain syndrome exercises, (n=20) Core stability group; Core stabilization and hip exercises will be given in addition to traditional patellofemoral pain syndrome exercises. (n=20) After obtaining the demographic information of the cases, before and after the treatment; Visual analog scale (VAS) change, Kuala scale change, Trunk forward flexion flexibility change, Hamstring muscle flexibility change, Sit-reach test change, Q angle measurement change, Normal joint movement change, McGill stabilization tests change, Timed get up and go test change, Single leg jump test change, Y balance test change, Muscle strength change will be evaluated by the same person using the Corbin Posture analysis change and Foot posture index (FPI) change parameters.

IMPLEMENTATION PROTOCOL

1. Control group; traditional patellofemoral pain syndrome exercises; isometric exercises 3 sets of 10 repetitions in one session, balance exercise 30/45 sec, one leg balance exercise 45/60 sec , stretching exercises 4 sets 5 repetitions 20 sec duration, off kinetic chain (CHC) AND open kinetic chain (ACZ) exercises were planned as 3 sets for 4 weeks and 3 days a week .
2. Core stability group; In addition to traditional patellofemoral pain syndrome exercises; hip muscle strengthening exercises are 3 sets of 10 repetitions in each session, and (core) stabilization exercises are 1st and 2nd weeks 2 sets 15 repetitions 3rd and 4th weeks 2 sets 5 repetition was planned for 4 weeks and 3 days a week.

While the patients will be exercised with a physiotherapist 1 day a week, the treatment will be followed as a home exercise program 2 days a week.

DETAILED DESCRIPTION:
SUBJECT AND OBJECTIVE OF THE RESEARCH The term patellofemoral pain syndrome (PFPS) is defined as retropatellar or peripatellar pain that occurs as a result of physical and biomechanical changes that causes pain in the anterior part of the knee related to changes in the patellofemoral joint.

Patellofemoral pain is one of the most common musculoskeletal problems, accounting for approximately 9-10% of all musculoskeletal complaints and 20-40% of all knee problems. PFPS is frequently encountered among young, physically active individuals. It is a common knee problem. It occurs most frequently in women, athletes and soldiers.

Many factors such as decrease in quadriceps femoris strength, decreased flexibility, activity mismatch between vastus medialis obliqua and vastus lateralis obliqua muscles, rotations between femur and tibia, excessive subtalar pronation, positional changes in the kneecap have been associated with patellofemoral pain syndrome. In a systematic analysis, it was observed that patients with PFPS had a decrease in the abduction/external rotation/extension strength of the affected side when compared to healthy individuals.

In a guideline regarding foot problems; It has been reported that foot pronation causes internal rotation of the tibia or femur (femoral anteversion), which disrupts the patellofemoral mechanism, while the pessary sergeant places more stress on the patellofemoral mechanism, especially when a person is running, since less softening and a harder contact are provided for the leg when the foot hits the ground.

In a controlled study involving patients with chronic PFPS, it was found that there was no significant difference between arthroscopy and home exercise program compared to home exercise alone, and home exercise alone was very effective.

The target in PFPS rehabilitation; to restore the functions of the joint and relieve pain. The first step in traditional rehabilitation is to strengthen the Quadriceps femoris (QF) and Vastus medialis obliqua (VMO) muscles. The treatment program consists of Open kinetic chain/Closed kinetic chain (ACZ/CHZ), stretching (iliotibial band, QF, hamstring, gastrocnemius, gastrocsoleus) exercises.

It was concluded that isokinetic exercises prevent extensor strength loss in patellofemoral pain syndrome, but they are not sufficient alone. In another study, it was found that hip strengthening exercises in addition to knee strengthening exercises were more effective in both improving function and reducing pain in sedentary women with PFPS than the group performing knee strengthening exercises alone. it was observed that the pain decreased more in the group in which both closed kinetic chain exercises and hip strengthening exercises were given compared to the group given only closed kinetic chain exercises.

In a randomized controlled study, core neuromuscular training was given in addition to routine physical therapy, and it was observed that patients improved more than routine physical therapy. In another study, core muscle strengthening exercises were given in addition to routine physical therapy and it was observed that it improved both pain and dynamic balance in patients compared to routine physical therapy alone.

Weight-bearing exercises are more functional than non-weight-bearing exercises because they require multi-joint movement, facilitate a functional muscle recruitment pattern, and stimulate proprioceptors. Because of these advantages, clinicians often recommend weight-bearing exercises in the rehabilitation of PFPS patients.

One systematic analysis determined the efficacy of physical exercise as a conservative treatment for patellofemoral pain syndrome by looking at the results of ten moderate to high quality clinical studies and showed that the most effective patellofemoral pain syndrome management included strengthening exercises for the hip at baseline. Due to their role in knee biomechanics, the addition of stretching exercises for the external rotator and abductor muscles, core muscles and proprioceptive, neuromuscular exercises " reduces pain in patellofemoral pain syndrome".

In the light of all these studies, when the literature was examined, very few studies were found that examined the effect of core stabilization exercises in individuals with patellofemoral pain syndrome, and these studies were only studied on certain parameters on women. The aim of this randomized controlled study; To investigate the multifactorial effectiveness of core stabilization exercises applied in patients diagnosed with patellofemoral pain syndrome.

Research Questions and Hypotheses:

What are the effects of core stabilization exercises in patellofemoral pain syndrome? H0: Core stabilization exercises are not effective on pain, functional level, balance, flexibility, muscle strength, normal joint movement, posture in patellofemoral pain syndrome.

H1: effective. Core stabilization exercises are effective on pain, functional level, balance, flexibility, muscle strength, normal joint movement and posture in patellofemoral pain syndrome.

Material and Method:

The study was planned as a randomized controlled trial. The number of volunteers to take part in the study was determined using the G-Power program. In the study, the randomized controlled study of 'Foroughi et al.' 45 named "Effects of Isolated Core Postural Control Training on Knee Pain and Function in Women with Patellofemoral Pain Syndrome: α=0.05, power 80% and effect size 0.3 were taken as an example. As a result of the calculations, it was found that there should be a total of 18 people, 9 people in each group. However, for a good statistical calculation or for the loss of cases, it was decided to take twice the result of this calculation. A total of 40 people, 20 people in each group, will be included in the study.

20/60 years old/with retropatellar pain that occurs during at least two of the activities and persists for at least one month While patients diagnosed with PFPS were included in the study; Patients with meniscus and ligament lesions , osteoarthritis , patellofemoral dislocation and/or subluxation history, osseous anomalies and history of knee surgery , pregnancy status, and patients using analgesics and anti-inflammatory drugs will not be included in the study.

Individuals will be divided into two groups by computerized randomization. Control group; Traditional patellofemoral pain syndrome exercises, (n=20) Core stability group; Core stabilization and hip exercises will be given in addition to traditional patellofemoral pain syndrome exercises. (n=20) After obtaining the demographic information of the cases change, before and after the treatment; Visual analog scale (VAS) change, Kuala scale change, Trunk forward flexion flexibility change, Hamstring muscle flexibility change, Sit-reach test change, Q angle measurement change, Normal joint movement change, McGill stabilization tests change, Timed get up and go test change, Single leg jump test change, Y balance test change, Muscle strength change will be evaluated by the same person using the Corbin Posture analysis change and Foot posture index (FPI) change parameters.

IMPLEMENTATION PROTOCOL

1. Control group; traditional patellofemoral pain syndrome exercises; isometric exercises 3 sets of 10 repetitions in one session, balance exercise 30/45 sec, one leg balance exercise 45/60 sec , stretching exercises 4 sets 5 repetitions 20 sec duration, off kinetic chain (CHC) AND open kinetic chain (ACZ) exercises were planned as 3 sets for 4 weeks and 3 days a week .
2. Core stability group; In addition to traditional patellofemoral pain syndrome exercises; hip muscle strengthening exercises are 3 sets of 10 repetitions in each session, and (core) stabilization exercises are 1st and 2nd weeks 2 sets 15 repetitions 3rd and 4th weeks 2 sets 5 repetition was planned for 4 weeks and 3 days a week.

While the patients will be exercised with a physiotherapist 1 day a week, the treatment will be followed as a home exercise program 2 days a week.

ELIGIBILITY:
Inclusion Criteria:

* 20/60 years old/with
* Occur during at least two activities of prolonged sitting, climbing stairs or inclines, squatting, running and jumping
* Retropatellar pain persisting for at least one month
* persons diagnosed with patellofemoral pain syndrome by the doctor are included in the study.

Exclusion Criteria:

* Meniscus and ligament lesions
* Osteoarthritis
* patellofemoral dislocation and/or subluxation history
* Osseous anomalies and history of knee surgery
* Pregnancy status
* Patients using analgesics and anti-inflammatory drugs will not be included.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
Demographic information form change | At baseline
  The patient's age, height, weight and disease history are questioned.
The visual analogue scale(VAS) change | Change from baseline the visual analogue scale at 4 weeks
  was described in a psychology journal in 1921. It is a visual scale, not a verbal one. This 11-point scale (from 0 to 10) has different names, but the verbal rating scale (VAS) is most often used. The VAS scoring has a 10 cm long straight line on which the patient can mark the degree of discomfort. For example, when measuring pain, you might have "no pain" on the left end of the line and "worst pain imaginable" on the right, or the like. The result can be read in millimeters (0 - 100 mm), or whole and half a centimeter (0 - 10 cm).
Kuala scale change | Change from baseline kuala scale at 4 weeks
  Kuala et al. He developed it in 1993 to assess subjective symptoms and functional limitations in PFPS. The score consists of 13 questions. These questions address activity-related pain when climbing stairs, squatting, running, jumping, performing weight-bearing activities, and sitting for long periods of time with the knee flexed. He also questions symptoms such as limping, swelling, patella subluxation, quadriceps muscle atrophy, lack of flexion, and flexion pain. The total score ranges from 0 to 100. A higher score indicates fewer complaints.
Y balance test change | Change from baseline Y balance test at 4 weeks
  The Y Balance test (YBT) is the most common dynamic balance assessment used in clinical practice and research to evaluate dynamic balance in 3 directions of reach YBT measures dynamic balance during single leg stance and requires strength, proprioception, and flexibility. YBT is a contralateral leg reaching system in one-leg stance anterior (ANT), posterolateral (PL), and posteromedial (PM) directions. A composite score is then calculated by summing the distance reached in 3 directions of reach (ANT, PL, and PM) relative to leg length. It has been reported that YBT predicts injury based on overall access performance (different threshold points depending on the sample) and asymmetry between the limbs (anterior access difference greater than 4 cm). In a study, YBT revealed inter-interpretive test-retest reliability and minimal measurement error.
Body front flexibility assessment change | Change from baseline Body front flexibility assessment at 4 weeks
  In this test, the person stands on a 15 cm high block and leans forward without bending the knees and tries to touch the fingertip. The test evaluates the flexibility of the lumbar region, hamstring muscles and M. gastrocnemius. The distance between the fingertip and the wooden block surface is measured with a tape measure, and the values that pass the block surface are recorded in cm as positive, and the values below the block surface as negative.
Muscle strength change | Change from baseline Muscle strength at 4 weeks
  Manual muscle testing does not consistently detect muscle strength deficiencies or clearly demonstrate the impact of such deficiencies on the knee. For this reason, functional performance testing may be preferred. Functional performance tests are a test for the knee and the entire lower extremity. 'Loudon et al.' He evaluated five different functional performance tests (anteromedial lunge, step-down, single-leg press, bilateral squat, balance reaching) in individuals with patellofemoral pain. All five of these tests revealed high reliability and correlated with changes in pain scales. Among these tests as muscle strength assessment in cases; anteromedial lunge, step down (step), balance reaching test will be used.
  If the patient cannot stabilize the pelvis by standing (on one leg) for 1 minute on the affected leg (the other side pelvis falls), it was decided to perform it on our patients, based on the study, which is said to be a sign of weakness of the hip muscles.
Normal joint movement change | Change from baseline Normal joint movement at 4 weeks
  Measurement will be made with G-Pro, an Android application. The G-Pro app is a highly accurate reliable tool for measuring knee flexion angle. Its results were found to be more significant and more accurate than the results of conventional instruments . It is preferred because it is easy to apply and has high reliability.
Corbin posture analyses change | Change from baseline Corbin posture analyses at 4 weeks
  Posture analyses will be performed to determine the changes in the posture of the individuals included in the study. These changes will be scored using the form prepared by Corbin et al. that includes lateral and posterior observations. This form is based on detecting postural disorders by observation made from the two planes mentioned and scoring them according to their severity. The scores will be added last and the postural status will be classified according to the total score. Postural anomalies were scored (0: none, 1: mild, 2: moderate, 3: severe). Postural scores obtained by looking from the lateral and posterior aspects are summed (0-2: excellent, 3-4: very good, 5-7: good, 8-11: moderate, 12≥ bad).
Foot Posture index or (FPI) change | Change from baseline Foot posture index at 4 weeks
  A six-item assessment scale (Foot Posture index or FPI) was developed in response to the need for a fast, easy and reliable method to measure foot position. The FPI consists of observing the bottom of the hind and forefoot of an individual standing in a relaxed position. The hindfoot is assessed by palpation of the talus head, observing the curves above and below the lateral malleoli, and inversion/eversion of the calcaneus. The forefoot consists of assessing the extent of abduction/adduction of the forefoot in the hindfoot, while checking the swelling in the talo-navicular joint area and the alignment of the medial longitudinal arch.
Assessment of hamstring muscle flexibility change | Change from baseline Assessment of hamstring muscle flexibility at 4 weeks
  In the supine position, the hip and knee are fixed in 90 degree flexion. The pivot point of the goniometer is placed on the lateral condyle of the femur. The knee angle will be measured by extending the patient's knee with the fixed arm parallel to the lateral midline of the femur and the mobile arm following the fibula. By subtracting the angular value found from 90 degrees, the shortness value will be obtained.
Sit and reach test change | Change from baseline Sıt and reach test at 4 weeks
  It was used for flexibility assessment. The patients will be asked to sit on the stretcher, with their legs extended and without shoes, and lean the soles of their feet on the front table. Then, the patient is asked to lie forward on the stretcher as much as possible, without flexing his knees, from his torso (waist and hip), and the extreme point where his fingers reach is cm. The best result will be recorded by measuring in terms of and repeating this test 3 times.
Q angle measurement change | Change from baseline Q angle measurement at 4 weeks
  It will be measured with a goniometer in the supine position, with the hip and knee extended. Between the line drawn from the spina iliaca anterior superior (SiAS) to the middle of the patella and the line drawn from the middle of the patella between the tuberositas tibia, this lateral angle will be measured 3 times and recorded. The average of the measurements will be recorded.
Mcgill stabilization tests change | Change from baseline Mcgill stabilization tests at 4 weeks
  Endurance tests known as McGill protocol; It was originally developed to evaluate core stabilization in patients with low back pain. This protocol consists of different endurance tests: lateral endurance, trunk flexor endurance, and trunk extensor endurance. In these tests, the time in seconds that the isometric posture is maintained is measured and recorded.
Timed start and go test change | Change from baseline Timed start and go test at 4 weeks
  The patients will be asked to start from a sitting position in a chair, get up with the given command, walk the predetermined distance of 3 meters as fast as they can, and return to their places. The time from the time they get up from the chair and sit down again will be recorded with the stopwatch. The measurements will be repeated 3 times and the average will be recorded in seconds.
Single leg jump test change | Change from baseline Single leg jump test at 4 weeks
  The patients begin the test in a position with their hands on their waists on one leg. Patients are asked to jump as far as possible in a parallel plane and land with the same leg. In the tape measure fixed to the ground, the distance between the patient's jump and the starting point is recorded in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Berrak VARHAN, Assoc. Prof., Study Director — Ethics committee protocol number 21-128
Locations (1):
- Istinye University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nunes GS, Stapait EL, Kirsten MH, de Noronha M, Santos GM. Clinical test for diagnosis of patellofemoral pain syndrome: Systematic review with meta-analysis. Phys Ther Sport. 2013 Feb;14(1):54-9. doi: 10.1016/j.ptsp.2012.11.003. Epub 2012 Dec 8. PMID 23232069
- [Background] Prins MR, van der Wurff P. Females with patellofemoral pain syndrome have weak hip muscles: a systematic review. Aust J Physiother. 2009;55(1):9-15. doi: 10.1016/s0004-9514(09)70055-8. PMID 19226237
- [Background] Tyler TF, Nicholas SJ, Mullaney MJ, McHugh MP. The role of hip muscle function in the treatment of patellofemoral pain syndrome. Am J Sports Med. 2006 Apr;34(4):630-6. doi: 10.1177/0363546505281808. Epub 2005 Dec 19. PMID 16365375
- [Background] Fredericson M, Yoon K. Physical examination and patellofemoral pain syndrome. Am J Phys Med Rehabil. 2006 Mar;85(3):234-43. doi: 10.1097/01.phm.0000200390.67408.f0. PMID 16505640
- [Background] Magalhaes E, Fukuda TY, Sacramento SN, Forgas A, Cohen M, Abdalla RJ. A comparison of hip strength between sedentary females with and without patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2010 Oct;40(10):641-7. doi: 10.2519/jospt.2010.3120. PMID 20508327
- [Background] Besier TF, Fredericson M, Gold GE, Beaupre GS, Delp SL. Knee muscle forces during walking and running in patellofemoral pain patients and pain-free controls. J Biomech. 2009 May 11;42(7):898-905. doi: 10.1016/j.jbiomech.2009.01.032. Epub 2009 Mar 6. PMID 19268945
- [Background] Steinberg N, Siev-Ner I, Peleg S, Dar G, Masharawi Y, Zeev A, Hershkovitz I. Joint range of motion and patellofemoral pain in dancers. Int J Sports Med. 2012 Jul;33(7):561-6. doi: 10.1055/s-0031-1301330. Epub 2012 May 4. PMID 22562733
- [Background] Tsuji T, Matsuyama Y, Goto M, Yimin Y, Sato K, Hasegawa Y, Ishiguro N. Knee-spine syndrome: correlation between sacral inclination and patellofemoral joint pain. J Orthop Sci. 2002;7(5):519-23. doi: 10.1007/s007760200092. PMID 12355123
- [Background] Juhn MS. Patellofemoral pain syndrome: a review and guidelines for treatment. Am Fam Physician. 1999 Nov 1;60(7):2012-22. PMID 10569504
- [Background] Noehren B, Hamill J, Davis I. Prospective evidence for a hip etiology in patellofemoral pain. Med Sci Sports Exerc. 2013 Jun;45(6):1120-4. doi: 10.1249/MSS.0b013e31828249d2. PMID 23274607
- [Background] Kettunen JA, Harilainen A, Sandelin J, Schlenzka D, Hietaniemi K, Seitsalo S, Malmivaara A, Kujala UM. Knee arthroscopy and exercise versus exercise only for chronic patellofemoral pain syndrome: a randomized controlled trial. BMC Med. 2007 Dec 13;5:38. doi: 10.1186/1741-7015-5-38. PMID 18078506
- [Background] Clijsen R, Fuchs J, Taeymans J. Effectiveness of exercise therapy in treatment of patients with patellofemoral pain syndrome: systematic review and meta-analysis. Phys Ther. 2014 Dec;94(12):1697-708. doi: 10.2522/ptj.20130310. Epub 2014 Jul 31. PMID 25082920
- [Background] Alaca R, Yilmaz B, Goktepe AS, Mohur H, Kalyon TA. Efficacy of isokinetic exercise on functional capacity and pain in patellofemoral pain syndrome. Am J Phys Med Rehabil. 2002 Nov;81(11):807-13. doi: 10.1097/00002060-200211000-00002. PMID 12394991
- [Background] Fukuda TY, Rossetto FM, Magalhaes E, Bryk FF, Lucareli PR, de Almeida Aparecida Carvalho N. Short-term effects of hip abductors and lateral rotators strengthening in females with patellofemoral pain syndrome: a randomized controlled clinical trial. J Orthop Sports Phys Ther. 2010 Nov;40(11):736-42. doi: 10.2519/jospt.2010.3246. PMID 21041965
- [Background] Ismail MM, Gamaleldein MH, Hassa KA. Closed kinetic chain exercises with or without additional hip strengthening exercises in management of patellofemoral pain syndrome: a randomized controlled trial. Eur J Phys Rehabil Med. 2013 Oct;49(5):687-98. Epub 2013 Jul 2. PMID 23820880
- [Background] Motealleh A, Mohamadi M, Moghadam MB, Nejati N, Arjang N, Ebrahimi N. Effects of Core Neuromuscular Training on Pain, Balance, and Functional Performance in Women With Patellofemoral Pain Syndrome: A Clinical Trial. J Chiropr Med. 2019 Mar;18(1):9-18. doi: 10.1016/j.jcm.2018.07.006. Epub 2019 Feb 10. PMID 31193229
- [Background] Chevidikunnan MF, Al Saif A, Gaowgzeh RA, Mamdouh KA. Effectiveness of core muscle strengthening for improving pain and dynamic balance among female patients with patellofemoral pain syndrome. J Phys Ther Sci. 2016 May;28(5):1518-23. doi: 10.1589/jpts.28.1518. Epub 2016 May 31. PMID 27313363
- [Background] Boling MC, Bolgla LA, Mattacola CG, Uhl TL, Hosey RG. Outcomes of a weight-bearing rehabilitation program for patients diagnosed with patellofemoral pain syndrome. Arch Phys Med Rehabil. 2006 Nov;87(11):1428-35. doi: 10.1016/j.apmr.2006.07.264. PMID 17084115
- [Background] Alba-Martin P, Gallego-Izquierdo T, Plaza-Manzano G, Romero-Franco N, Nunez-Nagy S, Pecos-Martin D. Effectiveness of therapeutic physical exercise in the treatment of patellofemoral pain syndrome: a systematic review. J Phys Ther Sci. 2015 Jul;27(7):2387-90. doi: 10.1589/jpts.27.2387. Epub 2015 Jul 22. PMID 26311988
- [Background] Rabelo ND, Lima B, Reis AC, Bley AS, Yi LC, Fukuda TY, Costa LO, Lucareli PR. Neuromuscular training and muscle strengthening in patients with patellofemoral pain syndrome: a protocol of randomized controlled trial. BMC Musculoskelet Disord. 2014 May 16;15:157. doi: 10.1186/1471-2474-15-157. PMID 24884455
- [Background] Song CY, Lin YF, Wei TC, Lin DH, Yen TY, Jan MH. Surplus value of hip adduction in leg-press exercise in patients with patellofemoral pain syndrome: a randomized controlled trial. Phys Ther. 2009 May;89(5):409-18. doi: 10.2522/ptj.20080195. Epub 2009 Mar 19. PMID 19299508
- [Background] Osteras B, Osteras H, Torstensen TA. Long-term effects of medical exercise therapy in patients with patellofemoral pain syndrome: results from a single-blinded randomized controlled trial with 12 months follow-up. Physiotherapy. 2013 Dec;99(4):311-6. doi: 10.1016/j.physio.2013.04.001. Epub 2013 Jun 10. PMID 23764516
- [Background] Moyano FR, Valenza MC, Martin LM, Caballero YC, Gonzalez-Jimenez E, Demet GV. Effectiveness of different exercises and stretching physiotherapy on pain and movement in patellofemoral pain syndrome: a randomized controlled trial. Clin Rehabil. 2013 May;27(5):409-17. doi: 10.1177/0269215512459277. Epub 2012 Oct 4. PMID 23036842
- [Background] Halabchi F, Mazaheri R, Mansournia MA, Hamedi Z. Additional Effects of an Individualized Risk Factor-Based Approach on Pain and the Function of Patients With Patellofemoral Pain Syndrome: A Randomized Controlled Trial. Clin J Sport Med. 2015 Nov;25(6):478-86. doi: 10.1097/JSM.0000000000000177. PMID 25654629
- [Background] Ummels PE, Lenssen AF, Barendrecht M, Beurskens AJ. Reliability of the Dutch translation of the Kujala Patellofemoral Score Questionnaire. Physiother Res Int. 2017 Jan;22(1). doi: 10.1002/pri.1649. Epub 2015 Aug 26. PMID 26308151
- [Background] Kuru T, Dereli EE, Yaliman A. Validity of the Turkish version of the Kujala patellofemoral score in patellofemoral pain syndrome. Acta Orthop Traumatol Turc. 2010;44(2):152-6. doi: 10.3944/AOTT.2010.2252. PMID 20676018
- [Background] Chimera NJ, Smith CA, Warren M. Injury history, sex, and performance on the functional movement screen and Y balance test. J Athl Train. 2015 May;50(5):475-85. doi: 10.4085/1062-6050-49.6.02. Epub 2015 Mar 11. PMID 25761134
- [Background] Engquist KD, Smith CA, Chimera NJ, Warren M. Performance Comparison of Student-Athletes and General College Students on the Functional Movement Screen and the Y Balance Test. J Strength Cond Res. 2015 Aug;29(8):2296-303. doi: 10.1519/JSC.0000000000000906. PMID 26203739
- [Background] Shaffer SW, Teyhen DS, Lorenson CL, Warren RL, Koreerat CM, Straseske CA, Childs JD. Y-balance test: a reliability study involving multiple raters. Mil Med. 2013 Nov;178(11):1264-70. doi: 10.7205/MILMED-D-13-00222. PMID 24183777
- [Background] Loudon JK, Wiesner D, Goist-Foley HL, Asjes C, Loudon KL. Intrarater Reliability of Functional Performance Tests for Subjects With Patellofemoral Pain Syndrome. J Athl Train. 2002 Sep;37(3):256-261. PMID 12937582
- [Background] Petersen W, Ellermann A, Gosele-Koppenburg A, Best R, Rembitzki IV, Bruggemann GP, Liebau C. Patellofemoral pain syndrome. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2264-74. doi: 10.1007/s00167-013-2759-6. Epub 2013 Nov 13. PMID 24221245
- [Background] Melian-Ortiz A, Varillas-Delgado D, Laguarta-Val S, Rodriguez-Aparicio I, Senent-Sansegundo N, Fernandez-Garcia M, Roger-de Ona I. [Reliability and concurrent validity of the app Goniometer Pro vs Universal Goniometer in the determination of passive knee flexion]. Acta Ortop Mex. 2019 Jan-Feb;33(1):18-23. Spanish. PMID 31480121
- [Background] Redmond AC, Crane YZ, Menz HB. Normative values for the Foot Posture Index. J Foot Ankle Res. 2008 Jul 31;1(1):6. doi: 10.1186/1757-1146-1-6. PMID 18822155
- [Background] Bliss LS, Teeple P. Core stability: the centerpiece of any training program. Curr Sports Med Rep. 2005 Jun;4(3):179-83. doi: 10.1007/s11932-005-0064-y. PMID 15907272
- [Background] Ferber R, Bolgla L, Earl-Boehm JE, Emery C, Hamstra-Wright K. Strengthening of the hip and core versus knee muscles for the treatment of patellofemoral pain: a multicenter randomized controlled trial. J Athl Train. 2015 Apr;50(4):366-77. doi: 10.4085/1062-6050-49.3.70. Epub 2014 Nov 3. PMID 25365133
- [Background] Foroughi F, Sobhani S, Yoosefinejad AK, Motealleh A. Added Value of Isolated Core Postural Control Training on Knee Pain and Function in Women With Patellofemoral Pain Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Feb;100(2):220-229. doi: 10.1016/j.apmr.2018.08.180. Epub 2018 Sep 26. PMID 30267667